CLINICAL TRIAL: NCT02188381
Title: The Role of Gut Microbiota in Hypertension: Brain-Gut Microbiome-Immune Axis in Hypertension
Brief Title: The Role of Gut Microbiota in Hypertension
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400233-N; 1R01HL132448-01 (NIH)
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2024-01

CONDITIONS: Hypertension
Keywords: Resistant Hypertension (RH); Uncontrolled Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Normal controls without hypertension: Control subjects will have a systolic BP <140mmHg with no cardiovascular disease. These subjects will provide a one time stool sample and a blood sample.
  Interventions: Other: Stool Sample and Blood Sample
- Controlled hypertension: Subjects with controlled hypertension will provide a one time stool sample and a blood sample.
  Interventions: Other: Stool Sample and Blood Sample
- Resistant hypertension: Resistant hypertension subjects will have systolic blood pressure (BP) ≥140 mmHg despite ≥3 anti-hypertensive medications of different classes. These subjects will provide a one time stool sample and a blood sample.
  Interventions: Other: Stool Sample and Blood Sample
- Prior enrolled in NCT 02133872: These subject will be asked to provide two stool samples and two blood samples. One at baseline and one after 3 months of therapy.
  Interventions: Other: Stool Sample and Blood Sample
- Remodeled Resistent Hypertension: Subjects with controlled hypertension will provide a one time stool sample and a blood sample.
  Interventions: Other: Stool Sample and Blood Sample

INTERVENTIONS:
Other: Stool Sample and Blood Sample — All subjects will provide a stool sample and a blood sample at baseline. Subjects in NCT02133872 will provide a second stool sample and blood sample at their 3 month visit.

SUMMARY:
Hypertension is the single most prevalent risk factor for heart diseases, heart failure, kidney failure and stroke. About 1 in 3 adults in the United States have hypertension. Approximately 28-30% of hypertensive patients suffer from resistant hypertension (RH). Inflammation has been implicated in the pathogenesis of the hypertension. Additional data suggests the involvement of gut microbiota in host normal cardiovascular functions and pathophysiology. Accumulating evidence demonstrates that antibiotic treatment benefits patients with acute coronary syndromes and reduces the incidence of ischemic cardiovascular events. Even though these studies did not address effects of antibiotic treatment on the gut microbiota, it is possible that gut microbiota could affect neurologic inflammation. Finally, intestinal microbiota has recently been proposed to modulate blood pressure (BP) through production of short-chain fatty acids. In order to investigate this, the investigators hypothesize that gut microbiota is involved in the neuroinflammation-mediated initiation and establishment of RH, and targeting gut microbiota by minocycline would produce beneficial outcomes in RH.

DETAILED DESCRIPTION:
This is a prospective cohort design. This study will enroll 388 subjects: 81 patients without HTN as a reference group, 81 patients with controlled HTN, 55 patients with uncontrolled HTN, 55 with remodeled RH, and 81 patients with RH to characterize gut microbiota composition. Subjects will provide stool samples for analysis. Subjects will also provide a blood sample for inflammatory marker and stem cell analysis.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and <80
* is competent and willing to provide consent

Inclusion criteria for each subject group:

* Control subjects will have a systolic BP <140mmHg with no cardiovascular disease
* Patients with controlled hypertension
* Patients with uncontrolled hypertension
* Resistant hypertension subjects will have systolic blood pressure (BP) ≥140 mmHg despite ≥3 anti-hypertensive medications of different classes one of which should be a diuretic
* Patients who are no longer RH subjects and have normal blood pressure
* Subjects participating in NCT 02133872 will be eligible to participate

Exclusion Criteria:

* currently pregnant or have been pregnant in the last 6 months;
* antibiotic treatment within 2 months of study enrollment;
* currently taking a medication (e.g., antibiotic, anti-inflammatory agents, glucocorticoids or other immune modulating medications);
* unwilling to discontinue vitamin or supplements, including probiotics, potentially affecting gut microbiota (vitamins/supplements and medications that possibly affect the gut microbiota should be discontinued for at least 2wks prior to stool collection);
* history of intestinal surgery, inflammatory bowel disease, celiac disease, lactose intolerance, chronic pancreatitis or other malabsorption disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will initially enroll 10 patients without hypertension as normal controls, and 10 patients with controlled hypertension and 10 patients with resistant hypertension to characterize gut microbiota. In addition, all patients enrolled in IRB# 102-2013 will be approached for possible participation.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Characterize gut microbiota composition at phylum level | 24 hours
  Stool samples to analyze the composition of the microbiota, extracted bacterial genomic DNA will be used as a template for PCR reactions targeting the V4-V5 variable regions of the 16S rRNA gene. Amplicons generated from the PCR will be run on the Illumina MiSeq sequencing platform available in our laboratory to profile microbial communities at phylum level.
Characterize gut microbiota composition at genus level | 24 hours
  Stool samples to analyze the composition of the microbiota, extracted bacterial genomic DNA will be used as a template for PCR reactions targeting the V4-V5 variable regions of the 16S rRNA gene. Amplicons generated from the PCR will be run on the Illumina MiSeq sequencing platform available in our laboratory to profile microbial communities at genus level.

SECONDARY OUTCOMES:
Reduction in BP is associated with changes in gut microbiota composition in RH subjects. | Baseline, 3 months
  Stool samples from patients enrolled in NCT 02133871 that received minocycline medication for resistant hypertension. Will be used to analyze the composition of the microbiota and data (taxonomic assignment) will be analyzed using QIIMEv1.3 pipeline to enumerate microbial population between samples derived from the cohorts.
IS hypertension associated with increased sympathetic activity and decreased parasympathetic activity and whether minocycline or other tetracyclines are effective to improve this balance | Baseline and 3 months
  Stool samples from patients enrolled in NCT 02133871 that received minocycline
To determine if characterization of gut microbiota in at risk patients predicts long term care utilization and/or cardiovascular outcomes | Up to 5 years
  Stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepline, MD, Principal Investigator — University of Florida
Locations (1):
- Cardiovascular Clinic at UF Health, Gainesville, Florida, United States